CLINICAL TRIAL: NCT00306423
Title: Rehabilitation Post Lumbar Microdiscectomy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Kornelia Kulig, Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #025027
Record Dates: First submitted 2006-03-21; First posted 2006-03-23 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Low Back Disorder
Keywords: exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor

INTERVENTIONS:
Procedure: Other: Exercise — exercise 3 times per week for 12 weeks
  Other Names: exercise 3 times per week for 12 weeks

SUMMARY:
The purpose of this study is to determine whether a rehabilitation program following lumbar microdiscectomy influences short-term (4 months) and long-term (up to 5 years)outcomes in quality of life, activity and endurance.

DETAILED DESCRIPTION:
Exercise

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years old
* Single level lumbar microdiscectomy

Exclusion Criteria:

* Potential subjects will be excluded is they exhibit symptoms suggestive of facet arthrosis or neurogenic claudication, or if their plain radiographs showed more than 50 percent loss of disc height at the relevant level.
* Patients in whom the protrusion occupied more than 50 percent of the sagittal diameter of the spinal canal or in whom sequestrated fragments were seen on MRI will also be excluded.

Other exclusion criteria will include:

* Previous back surgeries
* Presence of any other concurrent foot pathology besides leg and low back pain and associated single level disc injury
* Nervous system problems (e.g., stroke, dementia, seizures)
* Cognitive dysfunction (e.g. TBI, CVA, Alzheimer's)
* Uncontrolled cardiovascular disease
* Evidence of cord compression
* Uncontrolled hypertension
* Infection
* Severe respiratory disease
* Pregnancy
* Rheumatic joint disease
* Peripheral vascular disease with sensory loss of the foot
* Any condition that the subject identifies that might limit participation in physical activity

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2003-06 (Actual); Primary Completion 2011-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
ODI | pre and post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Kornelia Kulig, PhD, PT, Study Director — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States